CLINICAL TRIAL: NCT06331013
Title: CyberKnife Ultra-hypofractionated SBRT for Localized PROStatE cancEr With Dose-escalation to the Dominant Intraprostatic Lesion: is the Juice Worth the Squeeze? The PRO-SPEED Trial
Brief Title: CyberKnife Ultra-hypofractionated SBRT for Localized PROStatE cancEr
Acronym: PRO-SPEED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IEO 1872
Record Dates: First submitted 2024-03-13; First posted 2024-03-26 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CyberKnife SBRT treatment (Experimental): CyberKnife ultra-hypofractionated SBRT for localized Prostate cancer with dose-escalation to the dominant intraprostatic lesion
  Interventions: Radiation: CyberKnife ultra-hypofractionated SBRT

INTERVENTIONS:
Radiation: CyberKnife ultra-hypofractionated SBRT — CyberKnife ultra-hypofractionated SBRT for localized Prostate cancer with dose-escalation to the dominant intraprostatic lesion

SUMMARY:
This is a prospective observational study. The study will proceed with the enrollment of 60 patients in 2 years. he aim of the present study is to evaluate effectiveness of ultra-hypofractionated (UH) CyberKnife Stereotactic Body Radiation Therapy treatment on the whole prostate gland plus Simultaneous integrated boost (SIB) to the dominant intraprostatic lesions (DIL(s) in intermediate-unfavourable to high-risk Prostate Cancer (PCa) patients.

DETAILED DESCRIPTION:
The patient to be enrolled in the prospective observational phase will be screened at first visit; prescription of Prostate Specific Antigen (PSA) and testosterone analysis, uroflowmetry and multiparametric Magnetic Resonance Imaging (mpMRI) are mandatory if not already done.

Additional staging imaging (computed tomography (CT) and/or bone scan) will be required according to National Comprehensive Cancer Network (NCCN) category risk group.

Subsequently, for the eligible patient, the enrollment phase involves eco-guided transrectal insertion of 3-4 gold fiducials in the prostate gland.

CT with full bladder and empty rectum will be done after 7-10 days from fiducials insertion; CyberKnife-Stereotactic Body Radiation Therapy (SBRT) treatment will start after 5-7 days from the simulation CT. A total of 36.25 Gy to the prostate gland will be executed in 5 alternate days. For each treatment delivery, the patient is required to be prepared in roughly the same bladder and rectum filling condition of the simulation day. Finally, in the last treatment day QoL and both clinician- and patient-reported genitourinary (GU) and gastrointestinal (GI) acute toxicity assessment is required.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 and < 80 years
* Histologically confirmed adenocarcinoma of the prostate
* Low, Intermediate and high-risk category according to NCCN version 02.2021
* Clinically node negative and no distant metastasis
* Eastern Cooperative Oncology Group (ECOG) Performance Status <2
* Good urinary flow (peak flow >10 mL/s) or IPSS < 15
* Prostate volume < 100 cc
* Available mpMRI of the prostate
* Less than 3 DILs at mpMRI (if >2 DILs, only DILs with higher Prostate Imaging - Reporting and Data System (PIRADS) will be included and only PI-RADS >2)
* Written informed consent for treatment and research purpose

Exclusion Criteria:

* platelets count < 75000
* urethral stricture
* Previous pelvic RT
* Concomitant inflammatory bowel disease or other serious systemic comorbidities
* Previous prostatectomy
* Presence of hip prosthesis

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Acute GU and GI toxicities (RTOG) | 3 months
  Evaluation of acute genitourinary and gastrointestinal toxicity using Radiation Toxicity Grading (RTOG) distinguishing between lower toxicities (G1 and G2) and worse toxicities (G3 and G4)
Number of Participants with Late GU and GI toxicities (RTOG) | 24 months
  Evaluation of late genitourinary and gastrointestinal toxicity using Radiation Toxicity Grading (RTOG) distinguishing between lower toxicities (G1 and G2) and worse toxicities (G3 and G4)
Evaluation of patient-reported toxicity | 24 months
  Evaluation of patient-reported toxicity using International Prostatic Symptoms Score IPSS
Evaluation of patient-reported quality of life | 24 months
  Evaluation of patient-reported toxicity using International Index of Erectile Function Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Alicja Jereczek, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy